CLINICAL TRIAL: NCT00719251
Title: Effects of High Voltage Pulsed Current and Low Level Laser Therapy on Wound Healing in Diabetic Ulcers.
Brief Title: Effects of High Voltage Pulsed Current (HVPC) and Low Level Laser Therapy (LLLT) on Wound Healing in Diabetic Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Industrial de Santander (Other)
Responsible Party: Instituto Colombiano para el desarrollo de la ciencia y la tecnología - COLCIENCIAS, COLCIENCIAS
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1102-04-12916; 103-2003
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2009-03-05 (Estimated); Status verified 2009-03

CONDITIONS: Diabetic Foot Ulcer
Keywords: Complications of Diabetes Mellitus; Electric stimulation; Low-Level Laser Therapy
MeSH Terms: conditions — Diabetic Foot; Diabetes Complications | interventions — Electric Stimulation; Low-Level Light Therapy; Laser Therapy

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- HVG (Experimental): The patients received standard nursing care and HVPC
  Interventions: Device: High voltage pulsed current
- LG (Experimental): These patients received standard nursing care and LLLT
  Interventions: Device: Low level laser
- CG (Active Comparator): The control group only was treated with standard nursing care
  Interventions: Other: Standard nursing care

INTERVENTIONS:
Device: High voltage pulsed current — The patient´s wounds were treated for 45 minutes with HVPC three times a week for 16 weeks or until their ulcers closed. The active electrode made of aluminum foil was secured directly over the wound, which previously had been loosely packed with sterile gauze soaked with 0.9% saline solution. The dispersive electrode was placed 5 cms proximal to the wound.The electrical stimulator Intelect 340 stim model (Chattanooga Group) produces a twin peaked pulse and was applied with the following parameters: continuous mode, submotor level, 100 Hz pulse frequency and 100microseconds pulse duration. Prior to the beginning the study the electrical stimulator was calibrated with oscilloscope (Tektronix TDS 1002 model).
  Other Names: -electric stimulation; -high voltage stimulation
  Arms: HVG
Device: Low level laser — Wavelenght 633 nm (DMC - Brazil), power 30 mW, continuous, 2 J/cm2 in the edge of the ulcer and 1.5 J/cm2 in the bed, punctual application in direct contact, 3 times a week, 1 every alternate day, for 16 weeks or until the ulcer closed. The laser device was calibrated before each treatment session with a research radiometer (International Light).
  Other Names: Soft laser; Laser therapy; LLLT
  Arms: LG
Other: Standard nursing care — It was based to nursing intervention classification (NIC)46. These interventions were performed by a qualified nurse and included ulcer irrigation with physiological saline, sharp debridement as needed and maintenance of a moist wound environment with appropriate wound dressing. Patients were all educated regarding pressure off loading of the involved foot. All patients received standard wound care seven times a week for 16 weeks or until their ulcers closed.
  Other Names: Standard wound care; Wound care
  Arms: CG

SUMMARY:
The purpose of this study was to compare the effects of high voltage pulsed current and low level laser therapy on the healing process of diabetic foot ulcers.

DETAILED DESCRIPTION:
Based in the literature review we concluded that LLLT and HVPC are effective in the healing wound. We did not meet outcomes of previous clinical studies, where compare the effectivity of two physical technologies. For the high prevalence of diabetic foot ulcers, the amputation risk and the consequent impairment and dysfunction in the quality of life, and the associated high costs for this health problem, it is important that new studies that identified effective treatment alternatives for promoting wound closure.

ELIGIBILITY:
Inclusion Criteria:

* Ages 30 - 75 years
* Ulcer located on the legs or feet, stage I or II (Wagner Classification System)
* Diagnosis of diabetes mellitus according to World Health Organization criteria ( treatment with insulin or an oral hypoglycemic agent, two random glucose measurements major than 200 mg/dl, or a fasting glucose major than 140 mg/dl)

Exclusion Criteria:

* Uncontrolled diabetes
* Ulcer infection
* Lower limb amputation
* Orthopedic or neuromuscular pathologic conditions

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-03; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Characteristics of the wound | The wounds were evaluated at the beginning of the study (debridement previous), each two weeks during the intervention, at the finish of treatment and 30 and 60 days after completion of the intervention
Ankle Brachial Index (ABI) | The Ankle Braquial Index (ABI) was evaluated at the beginning of the study (debridement previous), each two weeks during the intervention, at the finish of treatment and 30 and 60 days after completion of the intervention.
Sensory testing with the Semmes-Weinstein monofilament | The monofilament testing was performed at the beginning and end of the treatment and 60 days thereafter.
Neuroconduction studies with the Nicolet Compass Meridian equipment. | The neuroconduction was performed at the beginning and end of the treatment and 60 days thereafter.
Quality of life with the EQ-5D. | The quality of life was applied at the begining and at the end of the treatment.

SECONDARY OUTCOMES:
Sociodemographic data like gender and age, were recorded. Additionally clinical history, deformities, alcohol dependence or smoking history, previous and present pharmacologic treatment and corticosteroids were included. | These outcome measures were assessed in the initial examination.

CONTACTS AND LOCATIONS:
Overall Officials: MARIA CRISTINA SANDOVAL ORTIZ, MSc in P.T., Principal Investigator — Industrial University of Santander; ESPERANZA HERRERA VILLABONA, M.Sc. Phys, Principal Investigator — Industrial University of Santander; DIANA MARINA CAMARGO LEMOS, M.Sc. Epid, Study Chair — Industrial University of Santander; RAFAEL CASTELLANOS, Dr., Study Chair — Industrial Universtiy of Santander
Locations (1):
- Industrial University of Santander UIS, Bucaramanga, Santander Department, Colombia

REFERENCES:
- [Background] Goldman RJ, Brewley BI, Golden MA. Electrotherapy reoxygenates inframalleolar ischemic wounds on diabetic patients: a case series. Adv Skin Wound Care. 2002 May-Jun;15(3):112-20. doi: 10.1097/00129334-200205000-00006. PMID 12055444
- [Background] Goldman R, Rosen M, Brewley B, Golden M. Electrotherapy promotes healing and microcirculation of infrapopliteal ischemic wounds: a prospective pilot study. Adv Skin Wound Care. 2004 Jul-Aug;17(6):284-94. doi: 10.1097/00129334-200407000-00010. PMID 15289715
- [Background] Peters EJ, Lavery LA, Armstrong DG, Fleischli JG. Electric stimulation as an adjunct to heal diabetic foot ulcers: a randomized clinical trial. Arch Phys Med Rehabil. 2001 Jun;82(6):721-5. doi: 10.1053/apmr.2001.23780. PMID 11387573
- [Background] Houghton PE, Kincaid CB, Lovell M, Campbell KE, Keast DH, Woodbury MG, Harris KA. Effect of electrical stimulation on chronic leg ulcer size and appearance. Phys Ther. 2003 Jan;83(1):17-28. PMID 12495409
- [Background] Hopkins JT, McLoda TA, Seegmiller JG, David Baxter G. Low-Level Laser Therapy Facilitates Superficial Wound Healing in Humans: A Triple-Blind, Sham-Controlled Study. J Athl Train. 2004 Sep;39(3):223-229. PMID 15496990
- [Background] Schindl A, Schindl M, Schon H, Knobler R, Havelec L, Schindl L. Low-intensity laser irradiation improves skin circulation in patients with diabetic microangiopathy. Diabetes Care. 1998 Apr;21(4):580-4. doi: 10.2337/diacare.21.4.580. PMID 9571346
- [Background] Demir H, Balay H, Kirnap M. A comparative study of the effects of electrical stimulation and laser treatment on experimental wound healing in rats. J Rehabil Res Dev. 2004 Mar;41(2):147-54. doi: 10.1682/jrrd.2004.02.0147. PMID 15558369
- [Background] Reddy GK. Comparison of the photostimulatory effects of visible He-Ne and infrared Ga-As lasers on healing impaired diabetic rat wounds. Lasers Surg Med. 2003;33(5):344-51. doi: 10.1002/lsm.10227. PMID 14677162
- [Background] Maiya GA, Kumar P, Rao L. Effect of low intensity helium-neon (He-Ne) laser irradiation on diabetic wound healing dynamics. Photomed Laser Surg. 2005 Apr;23(2):187-90. doi: 10.1089/pho.2005.23.187. PMID 15910184
- [Background] Al-Watban FA, Zhang XY, Andres BL. Low-level laser therapy enhances wound healing in diabetic rats: a comparison of different lasers. Photomed Laser Surg. 2007 Apr;25(2):72-7. doi: 10.1089/pho.2006.1094. PMID 17508840
- [Background] Zinman LH, Ngo M, Ng ET, Nwe KT, Gogov S, Bril V. Low-intensity laser therapy for painful symptoms of diabetic sensorimotor polyneuropathy: a controlled trial. Diabetes Care. 2004 Apr;27(4):921-4. doi: 10.2337/diacare.27.4.921. PMID 15047649
- [Background] Corazza AV, Jorge J, Kurachi C, Bagnato VS. Photobiomodulation on the angiogenesis of skin wounds in rats using different light sources. Photomed Laser Surg. 2007 Apr;25(2):102-6. doi: 10.1089/pho.2006.2011. PMID 17508845
- [Background] Silveira PC, Streck EL, Pinho RA. Evaluation of mitochondrial respiratory chain activity in wound healing by low-level laser therapy. J Photochem Photobiol B. 2007 Mar 1;86(3):279-82. doi: 10.1016/j.jphotobiol.2006.10.002. Epub 2006 Nov 20. PMID 17113781
- [Result] Kawalec, JS. Pfennigwerth, TC. Hetherington, VJ. Logan, JS. A review of lasers in healing diabetic ulcers. The foot. 14:68-71, 2004.
- See also: American Diabetes Association home page — http://www.diabetes.org
- See also: Universidad Industrial de Santander - home page — http://www.uis.edu.co/portal/english_version/english_version.html